CLINICAL TRIAL: NCT05755867
Title: Global Paroxysmal Nocturnal Hemoglobinuria (PNH) Patient Registry
Brief Title: Global PNH Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Aplastic Anemia and MDS International Foundation (Other)
Collaborators: National Organization for Rare Disorders (Other)
Responsible Party: Sponsor
Other Study IDs: AAMDSIF-PNH1
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Registry; Patient Registry; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PNH Patients: Individuals of any age with a confirmed diagnosis of PNH or diagnosis consistent with PNH are eligible for inclusion.

SUMMARY:
The primary aim of the Global Paroxysmal Nocturnal Hemoglobinuria (PNH) Patient Registry is to conduct a prospectively-planned and efficient natural history study that will result in a more comprehensive understanding of the disease and its course and pace over time. Other registry objectives include the following:

* Provide a convenient online platform for participants (or caregivers) to self-report cases of PNH.
* Develop a communications registry within the Global PNH Patient registry (e.g., to notify patients of research studies and clinical trials).
* Characterize and describe the Global PNH population as a whole, enhancing the understanding of disease prevalence and phenotype as well as the rate of progression of disease characteristics.
* Assist the PNH community with the development of recommendations and standards of care.
* Be a case-finding resource to be used for researchers who seek to study the pathophysiology of PNH, retrospectively collate intervention outcomes, and design prospective trials of novel treatments.

DETAILED DESCRIPTION:
The Global PNH Patient Registry is a prospective, longitudinal, web-based, observational natural history study. Participants with PNH will be followed throughout the course of their lives with either the participant or authorized respondents contributing data at varying intervals throughout the course of the study. Data will be collected at the start of the study (baseline), at least once per year or can be updated by the participant as needed. Data will be collected on demographics, quality of life, medical history, disease phenotypes, disease-related events, personal experience with PNH, general health status, medications, and diagnoses. The Global PNH Patient Registry provides a convenient online platform for participants; facilitates communication about PNH; gives researchers the ability to characterize the PNH population as a whole; assists the PNH community with the development of recommendations and standards of care and; and serves as a case-finding resource to be used for researchers to study the pathophysiology of PNH.

A Registry Advisory Board, that may include scientists, doctors, and patient advocates, will be assembled to oversee the conduct of the study. The Advisory Board will review aggregate registry data and the use of this registry, ensure proper evaluation of protocols requesting to use registry data and/or contact registry participants, and review any protocol or confidentiality deviations on a case- by by-case basis and ensure that any such deviations are reported to the IRB.

The registry will use a web-based interface to maximize accessibility to participants and clinicians world-wide. Following informed consent, participants will be invited to enter their data and information which will be stored indefinitely or until a participant revokes their consent to participate in the study. No experimental intervention is involved in participation in the Global PNH Patient registry study.

Annual maintenance will be funded by the Aplastic Anemia and MDS International Foundation (AAMDSIF) with support from industry partners. Registry participants will be automatically enrolled in NORD's Natural History Study Program (NHS), and their de-identified information aggregated with information from other rare diseases may be used for the purposes of cross disease analysis and cross-disease research to facilitate advocacy and further NORD's mission. De-identified information may be shared with other databases such as the Rare Disease Cures Accelerator-Data and Analytics Platform (RDCA-DAP). This will allow more researchers to use the information to do research.

ELIGIBILITY:
Inclusion Criteria:

- Individuals of any age with a confirmed diagnosis of PNH or diagnosis consistent with PNH are eligible for inclusion. PNH is defined as a genetic mutation in the PIG-A gene.

Individuals must be willing to provide informed consent. Participants can be:

* legal adult participants who are able to provide their own consent;
* children and adults unable to provide their own consent, for whom consent must be provided by a Legally Authorized Representative (LAR) who is a legal adult.
* Individuals must have at least periodic access to the internet and be able to comply with web-based study procedures and data collections

Exclusion Criteria:

* Individuals not able to read and understand English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age with a confirmed diagnosis of PNH or diagnosis consistent with PNH.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2031-05-06 (Estimated)

PRIMARY OUTCOMES:
Characterize and describe the Global PNH population | 5-10 years
  Understand disease prevalence and phenotype as well as the rate of progression of disease characteristics. Gather patient experiences including demographics, diagnostics, treatment, symptoms, and quality of life.

SECONDARY OUTCOMES:
Develop a communications registry | 5-10 years
  * Be a case-finding resource to be used for researchers who seek to study the pathophysiology of PNH, retrospectively collate intervention outcomes, and design prospective trials of novel treatments.
  * Notify patients of research studies and clinical trials as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Houk, MS, Principal Investigator — Aplastic Anemia and MDS International Foundation
Locations (1):
- Aplastic Anemia and MDS International Foundation, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that the Global PNH Patient Registry will be a valuable resource for current and future research. A Global PNH Patient Registry Advisory Board will ensure proper evaluation of protocols that request use of registry data and/or contact registry participants. To promote use of the repository, aggregate information about database contents will be updated quarterly or semi-annually and made available to the public. Such information may include number of registrants, prevalence of common diagnoses of registrants, demographic information, and percent willing to be contacted for future research. Investigators wanting to use the registry or contact participants will need to apply to the Advisory Board. The application will require information concerning: Principal Investigator, aims and hypotheses of the proposed research, where the research will be performed, and how the research will be funded.
Supporting Information: CSR
Time Frame: Data will be available 2 years after study start and will be analyzed through study ending.
Access Criteria: Sharing is subject to review by the Medical Advisory Committee

REFERENCES:
- See also: Description of the patient registry on the sponsor website — https://www.aamds.org/global-pnh-patient-registry
- See also: Link to registry platform where participants can enroll into the study — https://pnh.iamrare.org/